CLINICAL TRIAL: NCT01868451
Title: A Pilot Study of Brentuximab Vedotin Combined With AVD Chemotherapy in Patients With Newly Diagnosed Early Stage, Unfavorable Risk Hodgkin Lymphoma
Brief Title: Brentuximab Vedotin Combined With AVD Chemotherapy in Patients With Newly Diagnosed Early Stage, Unfavorable Risk Hodgkin Lymphoma
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Seagen Inc. (Industry); University of Rochester (Other); City of Hope Medical Center (Other); Stanford University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 13-034
Record Dates: First submitted 2013-05-30; First posted 2013-06-04 (Estimated); Last update posted 2025-07-09 (Actual); Status verified 2025-07

CONDITIONS: Hodgkin Lymphoma
Keywords: DACARBAZINE; DOXORUBICIN/ADRIAMYCIN; SGN-35 (BRENTUXIMAB VEDOTIN); VINBLASTINE; Involved-site radiation therapy (ISRT); Early stage; 13-034
MeSH Terms: conditions — Hodgkin Disease | interventions — Brentuximab Vedotin; Doxorubicin; Vinblastine; Dacarbazine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Cohort 1 (completed accrual) (Experimental): Patients received 4 cycles of brentuximab vedotin & AVD chemotherapy. Brentuximab vedotin, 1.2 mg/kg, will be administered on days 1 and 15 of each 28 day cycle. Doxorubicin 25 mg/m2, Vinblastine 6 mg/m2, & Dacarbazine 375 mg/m2 will be administered on days 1 and 15 of each 28 day cycle. This may be followed by 30 Gy involved site radiotherapy. Involved site radiotherapy should be initiated from 12 days to 42 days after completion of chemotherapy. It is mandatory to administer prophylactic growth factor support starting with cycle 1. Choice of growth factor and dosing can be determined at the discretion of the treating physican.
  Interventions: Drug: Brentuximab vedotin (SGN-35); Drug: Doxorubicin HCL; Drug: Vinblastine Sulfate; Drug: Dacarbazine; Radiation: Involved-Site Radiation Therapy (ISRT); Procedure: Interim PET
- Cohort 2 (Experimental): Patients with early stage, unfavorable risk Hodgkin lymphoma. The definition of disease bulk, one of the unfavorable risk features, has been updated, and is defined as the presence of any lymph node mass with transverse maximal diameter > 7.0 cm OR coronal maximal diameter > 7.0 cm. Patients will receive 4 cycles of brentuximab vedotin & AVD chemotherapy. Brentuximab vedotin, 1.2 mg/kg, will be administered on days 1 and 15 of each 28 day cycle. Doxorubicin 25 mg/m2, Vinblastine 6 mg/m2, and Dacarbazine 375 mg/m2 will be administered on days 1 & 15 of each 28 day cycle. This may be followed by 20 Gy involved site radiotherapy.
  Interventions: Drug: Brentuximab vedotin (SGN-35); Drug: Doxorubicin HCL; Drug: Vinblastine Sulfate; Drug: Dacarbazine; Radiation: Involved-Site Radiation Therapy (ISRT); Procedure: Interim PET
- Cohort 3 (Experimental): Patients will have early stage, unfavorable risk classical Hodgkin lymphoma with disease bulk defined as the presence of any lymph node mass with transverse maximal diameter > 7.0 cm or coronal maximal diameter > 7.0 cm. Patients will receive 4 cycles of brentuximab vedotin and AVD chemotherapy. Brentuximab vedotin, 1.2 mg/kg, will be administered on days 1 and 15 of each 28 day cycle. Doxorubicin 25 mg/m2, Vinblastine 6 mg/m2, and Dacarbazine 375 mg/m2 will be administered on days 1 and 15 of each 28 day cycle. This may be followed by 30.6 Gy CVRT.
  Interventions: Drug: Brentuximab vedotin (SGN-35); Drug: Doxorubicin HCL; Drug: Vinblastine Sulfate; Drug: Dacarbazine; Procedure: Interim PET; Radiation: consolidation volume RT (CVRT)
- Cohort 4 (Experimental): Patients will have early stage, unfavorable risk classical Hodgkin lymphoma with disease bulk defined as the presence of any lymph node mass with transverse maximal diameter > 7.0 cm or coronal maximal diameter > 7.0 cm. In this cohort. Pts will receive 4 cycles of brentuximab vedotin & AVD chemo. Brentuximab vedotin, 1.2 mg/kg, will be administered on days 1 & 15 of each 28 day cycle. Doxorubicin 25 mg/m2, Vinblastine 6 mg/m2, & Dacarbazine 375 mg/m2 will be administered on days 1 & 15 of each 28 day cycle. Pts whose PET scan is negative after 4 cycles of brentuximab vedotin & AVD chemotherapy will not receive RT. Pts whose PET scan is positive after 4 cycles of brentuximab vedotin & AVD chemo, but subsequent biopsy is neg, will also receive no RT. Upon MSK PI approval, if the simulation can't be covered by the institution or the pts insurance, a diagnostic IV contrast CT neck & diagnostic IV contrast CT CAP scan will be done in addition to the FDG-PET done after 4 cycles of chemo.
  Interventions: Drug: Brentuximab vedotin (SGN-35); Drug: Doxorubicin HCL; Drug: Vinblastine Sulfate; Drug: Dacarbazine; Procedure: Interim PET

INTERVENTIONS:
Drug: Brentuximab vedotin (SGN-35)
Drug: Doxorubicin HCL
Drug: Vinblastine Sulfate
Drug: Dacarbazine
Radiation: Involved-Site Radiation Therapy (ISRT)
  Arms: Cohort 1 (completed accrual); Cohort 2
Procedure: Interim PET
Radiation: consolidation volume RT (CVRT)
  Arms: Cohort 3

SUMMARY:
The purpose of this study is to compare the outcomes across the 4 different treatment groups. The investigators hope that this treatment will improve the ability to cure more patients with HL and also limit the long-term side effects from the treatment. Although eliminating radiation in cohort 4 will eliminate the risk for long-term side effects from radiation, it is also possible that with BV+AVD chemotherapy alone there may be an increased risk of the Hodgkin lymphoma coming back after initial treatment.

ELIGIBILITY:
Inclusion Criteria:

* Histologic diagnosis of classical, CD30 positive Hodgkin lymphoma confirmed at enrolling institution
* FDG-avid disease by FDG-PET/CT and measurable disease of at least 1.5 cm by CT
* Ann Arbor Stage I or II disease
* Disease bulk defined as any lymph node mass with transverse maximal diameter > 7.0 cm OR coronal maximal diameter > 7.0 cm on CT imaging
* Females of childbearing age must be on an acceptable form of birth control per institutional standards
* Ages 18 and over

Exclusion Criteria:

* Cardiac ejection fraction ≤ 50%
* Hemoglobin-adjusted diffusing capacity for carbon monoxide < 40%
* ANC≤1000/μl and Platelets≤75,000/μl
* Total bilirubin ≥ 2.0 mg/dl in the absence of a history of Gilbert's disease
* Serum creatinine clearance of <30 mL/min as estimated by the Cockcroft-Gault Method
* Known pregnancy or breast-feeding
* Known history of testing positive for human immunodeficiency virus (HIV) or known acquired immunodeficiency syndrome (AIDS)
* Medical illness unrelated to Hodgkin Lymphoma, which, in the opinion of the attending physician and/or MSKCC principal investigator, makes participation in this study inappropriate.
* Peripheral neuropathy > grade 1
* Patients receiving chronic treatment with systemic steroids. However, patients can receive up to 10 days of steroid therapy prior to starting treatment with BV+AVD.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 118 (Actual)
Dates: Start 2013-05 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
development of significant pulmonary toxicity | 1 year
  specifically non-infectious pneumonitis The definition of unacceptable pulmonary toxicity will be defined as the development of grade 2 or higher pneumonitis as defined by Common Terminology Criteria for Adverse Events (CTCAE version 4).
complete responses (all cohorts) | 1 year
  Evaluate the rate of PET-negative complete responses after completion of the treatment program (8 weeks (+/- 2 weeks) after completion of radiotherapy).

SECONDARY OUTCOMES:
Evaluate the prognostic significance | 1 year
  (i.e. correlation with progression free survival) of interim fluorodeoxyglucose-positron emission tomography (PET) in this patient population measured by visual analysis and semi-quantitative analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Anita Kumar, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (10):
- United States (10):
  - City of Hope, Duarte, California
  - Stanford University Medical Center, Stanford, California
  - Memorial Sloan Kettering Basking Ridge, Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth, Middletown, New Jersey
  - Memorial Sloan Kettering Bergen, Montvale, New Jersey
  - Memorial Sloan Kettering Commack, Commack, New York
  - Memorial Sloan Kettering Westchester, Harrison, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - University of Rochester Medical Center, Rochester, New York
  - Memorial Sloan Kettering Nassau, Uniondale, New York

REFERENCES:
- [Derived] Goldkuhle M, Kreuzberger N, von Tresckow B, Eichenauer DA, Specht L, Monsef I, Skoetz N. Chemotherapy alone versus chemotherapy plus radiotherapy for adults with early-stage Hodgkin's lymphoma. Cochrane Database Syst Rev. 2024 Dec 2;12(12):CD007110. doi: 10.1002/14651858.CD007110.pub4. PMID 39620432
- [Derived] Kumar A, Casulo C, Advani RH, Budde E, Barr PM, Batlevi CL, Caron P, Constine LS, Dandapani SV, Drill E, Drullinsky P, Friedberg JW, Grieve C, Hamilton A, Hamlin PA, Hoppe RT, Horwitz SM, Joseph A, Khan N, Laraque L, Matasar MJ, Moskowitz AJ, Noy A, Palomba ML, Schoder H, Straus DJ, Vemuri S, Yang J, Younes A, Zelenetz AD, Yahalom J, Moskowitz CH. Brentuximab Vedotin Combined With Chemotherapy in Patients With Newly Diagnosed Early-Stage, Unfavorable-Risk Hodgkin Lymphoma. J Clin Oncol. 2021 Jul 10;39(20):2257-2265. doi: 10.1200/JCO.21.00108. Epub 2021 Apr 28. PMID 33909449
- [Derived] Kumar A, Casulo C, Yahalom J, Schoder H, Barr PM, Caron P, Chiu A, Constine LS, Drullinsky P, Friedberg JW, Gerecitano JF, Hamilton A, Hamlin PA, Horwitz SM, Jacob AG, Matasar MJ, McArthur GN, McCall SJ, Moskowitz AJ, Noy A, Palomba ML, Portlock CS, Straus DJ, VanderEls N, Verwys SL, Yang J, Younes A, Zelenetz AD, Zhang Z, Moskowitz CH. Brentuximab vedotin and AVD followed by involved-site radiotherapy in early stage, unfavorable risk Hodgkin lymphoma. Blood. 2016 Sep 15;128(11):1458-64. doi: 10.1182/blood-2016-03-703470. Epub 2016 Jul 25. PMID 27458003
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/